CLINICAL TRIAL: NCT06554119
Title: Guangdong Provincial People's Hospital (Guangdong Academy of Medical Sciences), Southern Medical University
Brief Title: Surgical Treatments of Tricuspid Valve Regurgitation After Cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlei Huang, PhD, MD. pHD, Guangdong Provincial People's Hospital
Other Study IDs: Guangdong Provincial PHosp
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Tricuspid Valve Regurgitation; Complications, Longterm Outcome
Keywords: tricuspid valve regurgitation; technique advances; complications
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TVR: tricuspid valve replacement group，
  Interventions: Procedure: Huanlei Huang
- TVP: tricuspid valvuloplasty group
  Interventions: Procedure: Huanlei Huang

INTERVENTIONS:
Procedure: Huanlei Huang — tricuspid valve replacement or plasty

SUMMARY:
This study aims to present our center's experience in managing postoperative tricuspid valve regurgitation over the past 25years and to analyze the outcomes of these surgical treatments.

ELIGIBILITY:
Inclusion Criteria:patients who underwent surgical treatment from 1999 to 2023 for tricuspid valve disease following cardiac surgery

Exclusion Criteria: age <16，severe tricuspid regurgitation secondary to primary pulmonary hypertension, and those with substantial missing case data.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent surgical treatment from 1999 to 2023 for tricuspid valve disease following cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 1999-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
death rate | 1999-01 - 2025-01
  perioperative and longterm
complications | 1999-01 - 2025-01
  perioperative and longterm complications

SECONDARY OUTCOMES:
redo of tricuspid valve | 1999-01 - 2025-01
  redo of tricuspid valve during the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Huanlei Huang, Study Director — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital (Guangdong Academy of Medical Sciences), Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided